CLINICAL TRIAL: NCT03808558
Title: A Phase 2 Multi-center Pharmacodynamics Study of TVB-2640 in KRAS Mutant Non-small Cell Lung Carcinomas
Brief Title: Phase 2 Study of TVB-2640 in KRAS Non-Small Cell Lung Carcinomas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David E Gerber (Other)
Collaborators: Sagimet Biosciences Inc. (Industry); Cancer Prevention Research Institute of Texas (Other); Gateway for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, David E Gerber, PROFESSOR - Internal Medicine, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 022017-058
Record Dates: First submitted 2018-05-24; First posted 2019-01-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: KRAS Gene Mutation
MeSH Terms: interventions — TVB-2640

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TVB-2640 (Experimental): Patients will be administered TVB-2640 100mg/m2 orally once a day for 8 weeks.
  Interventions: Drug: TVB-2640

INTERVENTIONS:
Drug: TVB-2640 — TVB-2640 will be administered 100mg/m2 orally once a day for 8 weeks.

SUMMARY:
This is a prospective one-arm, two-stage phase 2 trial of TVB-2640 in KRAS mutant NSCLC patients. 13 patients will be treated with a minimum of 1 cycle of TVB-2640 therapy over 8 weeks.

DETAILED DESCRIPTION:
Patients with stable disease or partial/complete remissions will continue therapy.

The endpoints are response rate-RR, disease control rate-DCR, PFS-progression-free survival, CTCAEv5.0 toxicities, plasma lipid levels, collection of sebaceous secretion via Sebutape, and 11C-acetate PET tumor imaging.

In the first stage, 13 patients will be enrolled. If fewer than 2 patients achieve response, the study will be stopped. If 2 or more patients have a radiographic response, an additional 21 patients will be enrolled , for a total accrual of 34 patients.

ELIGIBILITY:
Inclusion:

1. Metastatic or advanced stage, histologically or cytologically confirmed NSCLC and molecular identification of oncogenic KRAS mutation.

   * KRAS mutant NSCLC must be refractory, relapsed, and previously treated with doublet chemotherapy and immune checkpoint inhibitor (unless there is a specific contraindication to checkpoint inhibitor).
   * Molecular characterization (tissue- or blood-based [ie, cell-free/circulating tumor DNA]) must have been performed and must have demonstrated an oncogenic KRAS mutation (e.g., exon 12, 13, 61, or 117 mutation detected by sequencing) by a CLIA-certified assay (source documentation required). KRAS mutations at other codons require review and approval by Study Chair.
2. Subjects' EGFR mutation and ALK gene rearrangement status must be known prior to study entry. Subjects with EGFR mutation or ALK gene rearrangement must have progressed after appropriate FDA-approved targeted therapy options prior to eligibility.
3. Patient has evidence of disease progression on most recent line of therapy.
4. Patient has measurable disease by RECIST v1.1 (Eisenhauer, 2009).
5. Age ≥ 18 years.
6. ECOG performance status of 0 or 1.
7. Predicted life expectancy of >3 months.
8. Adequate organ and marrow function as defined below:

   * absolute neutrophil count ≥ 1,500/mcL
   * platelets ≥ 75,000/mcL
   * total bilirubin <2X institutional upper limit of normal
   * AST and ALT ≤5X institutional upper limit of normal
   * serum creatinine <1.5X institutional upper limit of normal
   * LVEF >50%
   * QTcF <470msec
9. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

     * Has not undergone a hysterectomy or bilateral oophorectomy; or
     * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
10. No significant ischemic heart disease or myocardial infarction within 6 months of first dose of TVB-2640 and with current adequate cardiac function as in 3.1.8.
11. Ability to understand and the willingness to sign a written informed consent.

Exclusion:

1. Patient is unable to swallow oral medications or has impairment of GI function or GI disease that may significantly alter drug absorption such as active inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome.
2. Patient has a history of risk factors for torsade de pointes such as uncontrolled heart failure, severe hypokalemia with potassium less than 3mM/L, history of long QT syndrome or require use during study participation of concomitant medications known to prolong QT/QTc interval.
3. Patients who require use of strong CYP3A4/5 agonists or inhibitors during study participation.
4. Patient has uncontrolled or severe intercurrent medical condition including uncontrolled brain metastases. Patients with stable brain metastases either treated or untreated, on a stable dose of steroids/anticonvulsants, with no dose increase within 4 weeks before the first dose of TVB-2640, and no anticipated dose change, are allowed.
5. Patient underwent major surgery within 4 weeks before the first dose of TVB-2640 or received cancer-directed therapy either chemotherapy, radiotherapy, hormonal therapy, biologic or immunotherapy, etc. or an investigational drug or device within 2 weeks (6 weeks for mitomycin C and nitrosoureas) or 5 half-lives of that agent, whichever is shorter before the first dose of TVB-2640. In addition, any drug- related toxicity, with the exception of alopecia, an endocrinopathy controlled with replacement therapy, or a clinically stable toxicity not expected to increase from study therapy (eg, cisplatin-associated ototoxicity) should have recovered to <Grade 1.
6. If female, patient is pregnant or breast-feeding.
7. Patient has evidence of a serious active infection-infection requiring treatment with intravenous antibiotics.
8. Patient has known immunodeficiency virus-HIV or hepatitis B or C infection, as such patients may be at increased risk for toxicity due to concomitant treatment and disease-related symptoms may preclude accurate assessment of the safety of TVB-2640.
9. Patient has an important medical illness or abnormal laboratory finding that, in the Investigator's opinion, would increase the risk of participating in this study.
10. Patients with prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational agent.
11. History of clinically significant dry eye (xerophthalmia) or other corneal abnormality or, if a contact lens wearer, does not agree to abstain from contact lens use from baseline through the last study drug dose.
12. Patient has a known allergy or hypersensitivity to components of TVB-2640.
13. Patient has a prior history of hypersensitivity, drug/radiation-induced, or other immune-mediated pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate of TVB-2640 | every 8 weeks through study completion, an average of 1 year
  Determine Disease control rate of TVB-2640 in KRAS mutant NSCLC patients through RECIST and toxicity profile.
Response rate of TVB-2640 | every 8 weeks through study completion, an average of 1 year
  Determine response rate of TVB-2640 in KRAS mutant NSCLC patients through RECIST and toxicity profile.

SECONDARY OUTCOMES:
Safety profile of TVB-2640 | Pretreatment and four weeks of treatment.
  Secondary endpoints are 11C-acetate tumor uptake pretreatment and at four weeks of treatment and plasma lipidomics pretreatment and at four weeks of treatment.
Establish the predictive value of 11C-acetate PET | Pretreatment and four weeks of treatment.
  To establish the predictive value of 11C-acetate PET pretreatment and post-treatment tumor uptake for disease control rate and response rate
Mean change in fasting plasma lipidomics | Pretreatment and four weeks of treatment.
  Blood samples for fasting plasma lipidomics will be collected at baseline and four weeks of treatment.
Mean change in sebaceous secretion of fatty acids | Pretreatment and four weeks of treatment.
  Sebutabe collection of sebaceous secretion of fatty acids will be performed at baseline and four weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Gerber, MD, Principal Investigator — Professor
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No